CLINICAL TRIAL: NCT06182943
Title: Clinical Evaluation of Surrounding Electroacupuncture in the Treatment of Acute Lateral Ankle Sprain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Hu Qimiao, lecturer, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSLL-ZN-2023-011-01
Record Dates: First submitted 2023-12-01; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electroacupuncture group (Experimental): electroacupuncture combined with surrounding acupuncture
  Interventions: Other: electroacupuncture combined with surrounding acupuncture
- sham electroacupuncture group (Sham Comparator): sham electroacupuncture
  Interventions: Other: sham electroacupuncture
- ice compress combined with brake rest group (Placebo Comparator): ice compress combined with brake rest
  Interventions: Other: ice compress combined with brake rest

INTERVENTIONS:
Other: electroacupuncture combined with surrounding acupuncture — electroacupuncture combined with surrounding acupuncture
  Arms: electroacupuncture group
Other: sham electroacupuncture — sham electroacupuncture
  Arms: sham electroacupuncture group
Other: ice compress combined with brake rest — ice compress combined with brake rest
  Arms: ice compress combined with brake rest group

SUMMARY:
Comparison and evaluation of the difference in clinical efficacy of electroacupuncture combined with surrounding acupuncture and sham electroacupuncture groups and control group (ice compress combined with brake rest group) in the treatment of ALAS by means of musculoskeletal ultrasound technique.

DETAILED DESCRIPTION:
1. To evaluate the efficacy and safety of electroacupuncture combined with surrounding acupuncture in the treatment of ALAS,and compare its differences and advantages with traditional therapy.
2. To investigate the effect of electroacupuncture combined with surrounding acupuncture on the physiological and biochemical changes of the affected nerve,muscle and ligament, as well as its mechanism and pathway.
3. To investigate the influence of treatment time,frequency,intensity,stimulation point and other factors on the therapeutic effect and mechanism,further optimize the treatment plan and improve the therapeutic effect and efficiency.
4. To demonstrate the unique advantages and value of acupuncture analgesia,strengthen the concept and practice of integrated Chinese and Western medicine,and make contributions to promoting the application and development of acupuncture analgesia in the field of orthopedics and traumatology.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for a grade I or II injury;
* Onset time≤48h;
* The patient aged between18 and 60, gender is not limited;
* The skin of the ankle joint on the affected side is intact, without breakage or ulceration;

Exclusion Criteria:

* Combined with ankle fracture;
* Grade III injury or complete ligament rupture;
* Those who cannot comply with the treatment program. Those with keloid, localized combination of other skin diseases, and those who are not suitable for electroacupuncture treatment;
* Those with serious cardiovascular, cerebrovascular, hepatic, renal, hematopoietic system or systemic failure, connective tissue disease, hemophilia, diabetes mellitus, malignant tumors, and those who are prone to bleeding tendency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Kofoed | before treatment（baseline,week0）, after treatment(week4) and 1 week after treatment（follow-up,week5）.
  The Kofoed evaluation system was divided into 3 items, which were evaluated before treatment, 3 weeks after treatment and after treatment. The ankle joint function was evaluated mainly from three aspects of pain, function and range of motion, with a total score of 100.

SECONDARY OUTCOMES:
musculoskeletal ultrasound quantitative measurement | before（baseline,week0）and after treatment(week4).
  The thickness of lateral collateral ligament of ankle joint was measured by GE LOGIQ-e portable color Doppler ultrasonography before and after treatment. The frequency of linear array probe was 8 ~ 12 mHz.
circumference of ankle joint | before treatment（baseline,week0）, after treatment(week4) and 1 week after treatment（follow-up,week5）.
  The circumference of ankle joint was measured in 3 groups before, 3 weeks and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xianming Lin, Phd, Study Chair — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China